CLINICAL TRIAL: NCT01764321
Title: A Multi-center, Noninterventional Study With Certolizumab Pegol in Comparison With Any Other Subcutaneous TNF Inhibitor in Two Parallel Groups in Biologic Naive Patients With Rheumatoid Arthritis
Brief Title: Noninterventional Examination of Subcutaneous (sc) Tumor Necrosis Factor (TNF) Inhibitors
Acronym: NexT
Status: Completed | Type: Observational
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: RA0097
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol; Cimzia®; TNF inhibitor; DMARD; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Certolizumab Pegol treatment: Certolizumab Pegol in combination with at least one Disease Modifying Antirheumatic Drug (DMARD)
- Other Tumor Necrosis Factor TNF inhibitor treatment: Other subcutaneous (sc) Tumor Necrosis Factor (TNF) inhibitor (Adalimumab, Golimumab, Etanercept) in combination with at least one Disease Modifying Antirheumatic Drug (DMARD)

SUMMARY:
This prospective, post marketing, observational, Noninterventional Study (NIS) is designed to compare drug persistence in patients treated with Certolizumab Pegol (CZP) and patients treated with any other subcutaneously (sc) administered Tumor Necrosis Factor (TNF) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA)
* Moderate to severe disease activity of RA
* The patient receives Tumor Necrosis Factor (TNF) inhibitor in combination with at least 1 synthetic Disease Modifying Antirheumatic Drug (DMARD)
* The decision to prescribe a TNF inhibitor in combination with DMARD is made by the treating physician, prior to and independently from the decision to include the patient in this Non-Interventional Study (NIS)
* Male or female patients ≥ 18 years of age, considered by the treating physician to be reliable and capable of adhering to the observational plan (eg, able to understand and complete questionnaires)
* The patient personally signed and dated Patient Data Consent Form (PDCF) prior to Visit 2
* Treatment is according to the Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* Known contraindications to Tumor Necrosis Factor (TNF) inhibitors
* Prior use of any TNF inhibitors (including Adalimumab, Etanercept, Infliximab, Certolizumab, or Golimumab), or other biologic DMARDs (including Abatacept, Rituximab, Tocilizumab, or Anakinra)
* Participation in an investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed Rheumatoid Arthritis (RA)
Sampling Method: Non-Probability Sample
Enrollment: 1723 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients demonstrating persistence to the initially prescribed Tumor Necrosis Factor (TNF) inhibitor after 24 months of treatment | up to Week 104
  For a patient to be classified as persistent he or she must be classified as an early responder up to Week 12 and be continuously treated up to Week 104 with the initially prescribed Tumor Necrosis Factor (TNF) inhibitor at a dose not greater than that initially prescribed according to the Summary of Product Characteristics (SmPC).
  For the definition of persistence rate for the primary variable, patients will be classified as early responders if their Disease Activity Score 28 (DAS28) shows a reduction of >=1.2 from Baseline or decreases to <=3.2 (Low Disease Activity (LDA) or remission) up to Week 12.
  Non responders up to Week 12 will be counted as non persistent to the initially prescribed TNF inhibitor treatment.
  Patients who stop the initially prescribed TNF inhibitor treatment will not be counted as persistent, except if treatment with TNF inhibitor is stopped because the patient is in clinical remission.

SECONDARY OUTCOMES:
Proportion of patients achieving early clinical response to treatment based on Disease Activity Score 28 (DAS28) reduction of ≥ 1.2 or DAS28 decrease to ≤ 3.2 up to Week 12 | From Baseline up to Week 12
Proportion of patients achieving early clinical response to treatment based on DAS28 reduction of ≥ 1.2 or DAS28 decrease to ≤ 3.2, and being in DAS28 remission (DAS28<2.6) or ([LDA] DAS28<=3.2) at Week 104 | From Baseline up to Week 12 and to Week 104
  * LDA is defined as DAS28 ≤ 3.2
  * DAS28 is defined as Disease Activity Score 28
Proportion of patients not achieving early clinical response to treatment based on DAS28 reduction of >=1.2 or DAS28 decrease to <=3.2, and being in DAS28 remission (DAS28<2.6) or LDA (DAS28<=3.2) at Week 104 | From Baseline up to Week 12 and to Week 104
  * LDA is defined as DAS28 ≤ 3.2
  * DAS28 is defined as Disease Activity Score 28
Proportion of patients achieving early clinical response to treatment based on Disease Activity Score 28 (DAS28) reduction of ≥ 1.2 up to Week 12 | From Baseline up to Week 12
Proportion of patients achieving early clinical response to treatment based on Disease Activity Score 28 (DAS28) reduction of ≥ 1.2, and being in DAS28 remission (DAS28<2.6) or LDA (DAS28<=3.2) at Week 104 | From Baseline up to Week 12 and to Week 104
  Low Disease Activity (LDA) is defined as DAS28 ≤ 3.2
Proportion of patients not achieving early clinical response to treatment based on DAS28 reduction of >=1.2, and being in DAS28 remission (DAS28<2.6) or LDA (DAS28<=3.2) at Week 104 | From Baseline up to Week 12 and to Week 104
  Low Disease Activity (LDA) is defined as DAS28 ≤ 3.2
Proportion of patients who discontinued the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to lack/loss of efficacy during the duration of the study (up to Week 104) | From Baseline up to Week 104
Proportion of patients who discontinued the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to Adverse Events (AEs) during the duration of the study (up to Week 104) | From Baseline up to Week 104
Proportion of patients who discontinued the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to any other reasons during the duration of the study (up to Week 104) | From Baseline up to Week 104
Time to discontinuation of the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment at the dose recommended according to the Summary of Product Characteristics (SmPC) during the duration of the study | From Baseline up to Week 104
Time to discontinuation of the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to lack/loss of efficacy during the duration of the study (up to Week 104) | From Baseline up to Week 104
Time to discontinuation of the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to Adverse Events (AEs) during the duration of the study (up to Week 104) | From Baseline up to Week 104
Time to discontinuation of the initially prescribed Tumor Necrosis Factor (TNF) inhibitor treatment due to any other reasons during the duration of the study (up to Week 104) | From Baseline up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (122):
- Germany (122):
  - 039, Aachen
  - 079, Aachen
  - 017, Altenburg
  - 044, Altenholz
  - 082, Amberg
  - 030, Bad Bramstedt
  - 073, Bad Doberan
  - 134, Bad Homburg
  - 010, Bad Kreuznach
  - 153, Bad Kreuznach
  - 023, Bad Nauheim
  - 132, Bad Neuenahr-Ahrweiler
  - 196, Bad Pyrmont
  - 046, Bautzen
  - 125, Bautzen
  - 031, Bayreuth
  - 033, Bayreuth
  - 018, Berlin
  - 019, Berlin
  - 036, Berlin
  - 040, Berlin
  - 058, Berlin
  - 072, Berlin
  - 087, Berlin
  - 099, Berlin
  - 100, Berlin
  - 101, Berlin
  - 005, Bochum
  - 194, Braunschweig
  - 021, Burghausen
  - 179, Chemnitz
  - 075, Cottbus
  - 027, Darmstadt
  - 062, Donaueschingen
  - 089, Dresden
  - 110, Dresden
  - 063, Düsseldorf
  - 014, Elmshorn
  - 080, Erfurt
  - 142, Erlangen
  - 176, Essen
  - 008, Frankenberg
  - 016, Frankfurt
  - 098, Frankfurt
  - 054, Freiberg
  - 041, Freiburg im Breisgau
  - 147, Freiburg im Breisgau
  - 188, Friedrichroda
  - 140, Geilenkirchen
  - 164, Geislingen an der Steige
  - 133, Giessen
  - 191, Giessen
  - 143, Goslar
  - 032, Göttingen
  - 025, Greifswald
  - 029, Halle
  - 186, Halle
  - 002, Hamburg
  - 006, Hamburg
  - 052, Hamburg
  - 056, Hamburg
  - 070, Hamburg
  - 107, Hanover
  - 136, Hanover
  - 048, Heidelberg
  - 057, Heidelberg
  - 124, Herne
  - 043, Hildesheim
  - 053, Hofheim
  - 092, Hoyerswerda
  - 096, Jena
  - 180, Karlsruhe
  - 184, Kronach
  - 004, Leipzig
  - 068, Leipzig
  - 013, Ludwigsfelde
  - 114, Lübeck
  - 034, Magdeburg
  - 177, Mainz
  - 195, Mansfeld
  - 028, Marktredwitz
  - 049, Mittelherwigsdorf
  - 055, Mönchengladbach
  - 015, München
  - 020, München
  - 093, München
  - 111, München
  - 175, München
  - 037, Naunhof
  - 047, Neubrandenburg
  - 078, Neuss
  - 090, Neuss
  - 109, Nienburg
  - 076, Offenburg
  - 035, Planegg
  - 097, Plauen
  - 051, Potsdam
  - 187, Potsdam
  - 061, Püttlingen
  - 185, Radebeul
  - 123, Rendsburg
  - 118, Rostock
  - 112, Saarbrücken
  - 121, Schwerin
  - 122, Schwerin
  - 144, Schwerin
  - 193, Seesen
  - 115, Stadtbergen
  - 171, Stolberg
  - 074, Stuttgart
  - 146, Stuttgart
  - 085, Traunstein
  - 152, Treuenbrietzen
  - 009, Tübingen
  - 059, Tübingen
  - 077, Weener
  - 113, Winsen
  - 065, Wuppertal
  - 106, Würselen
  - 042, Würzburg
  - 182, Zwickau
  - 001, Zwiesel